CLINICAL TRIAL: NCT00190021
Title: Donepezil as Add-On Treatment of Psychotic Symptoms in Patients With Dementia of the Alzheimer's Type
Brief Title: Donepezil Treatment of Psychotic Symptoms in Dementia Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beersheva Mental Health Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMHC-3495CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2005-10

CONDITIONS: Dementia of Alzheimer Type
Keywords: Alzheimer's type dementia; donepezil; double-blind
MeSH Terms: interventions — Donepezil

INTERVENTIONS:
Drug: donepezil

SUMMARY:
Conventional psychotropic medications may be used to treat behavioral disturbances and psychotic symptoms in patients with dementia and they are the drugs of choice for treating delusions and hallucinations. However the sensitivity to side effects in these patients often restricts the use of these agents (2, 3). Although, atypical antipsychotics have some advantages compared with conventional neuroleptics, they also are associated with side effects (5, 6).

Cholinesterase inhibitors (ChEIs) enhance neuronal transmission by increasing the availability of acetylcholine in muscarinic and nicotinic receptors. According to findings of some researchers ChEIs have psychotropic effects and may play an important role in controlling neuropsychiatric and behavioral disturbances in patients with Alzheimer's disease (7-10). These agents may also contribute to the management of other disorders with cholinergic system abnormalities and neuropsychiatric symptoms such as visual hallucinations (11).

Donepezil is a piperidine-based reversible, noncompetitive ChEI, which is indicated in the management of patients with Alzheimer's disease of mild to moderate severity (12-14). Preliminary observations suggest the possible value of ChEIs in the amelioration of psychotic symptoms in patients with dementia of the Alzheimer's type (DAT), dementia with Lewy bodies and patients suffering from Parkinson's disease (11-18).

The results of our study (18) indicate that the addition of donepezil to perphenazine resulted in qualitatively superior clinical gains compared to higher doses of neuroleptic therapy without donepezil.

The finding of the pilot study although impressive, stem from data regarding a rather small sample. The present (second) phase of the study will include a larger sample of patients. We now intend to examine 80 inpatients, aged 65-90 years old, suffering from DAT.

DETAILED DESCRIPTION:
Criteria for inclusion into the study will be: 1) DSM-IV diagnosis of Dementia of the Alzheimer type with psychotic symptoms such as hallucinations and delusions, aggression/agitation, irritability, and disinhibition that called for the administration of antipsychotic drugs; 2) duration of psychotic symptoms at least 2 weeks before beginning of treatment; 3) lack of improvement of psychotic symptoms (less than 25% on Positive and Negative Symptoms Scale (PANSS) during perphenazine treatment (8 mg/day) for at least three weeks; 4) drug regimen for physical disease of all patients was unchanged for at least three months before the study.

Exclusion criteria include: 1) a vascular dementia; 2) concurrent Axis I DSM-IV diagnoses (delirium, schizophrenia, delusional disorders, and affective disorders) 3) significant medical illness (cardiovascular, liver, renal, endocrinal, vitamin B12 or folic acid deficiency, and neurological illnesses); 4) drug or/and alcohol addiction.

The study design will be a double blind group study, lasting for 9 weeks. Complete physical and laboratory examinations will be performed on all inpatients. Subjects will be randomized in a 1:1 fashion to receive treatment with 4 mg of perphenazine or 5 mg of donepezil or placebo in addition to the perphenazine treatment (8 mg/day) that they have received for the past 3 weeks (baseline). According to mental state (improvement less than 20% on PANSS scores), perphenazine dose will be elevated by 4 mg/day to maximum 16 mg/day in the first group, and donepezil dose will be increased by 5 mg/day to maximum 10 mg/day in the second group) and placebo will be elevated up to 2 capsules/day in the third group. All preparations will be administered in identical capsules made by a professional pharmacist, and supplied in individual number-coded packages.

Assessments for psychotic symptoms will be done using PANSS and CGI at baseline and repeated weekly. Assessments for extrapyramidal side effects will be done using AIMS at baseline and repeated every week. In addition, both at the beginning and at the end of the study, all patients will be assessed with MMSE and GDS. Complete blood profiles, and urine analysis will be performed at screening and at week 9.

References

1. Evans DA. Estimated prevalence of Alzheimer's disease in the United States. Milbank Q 1990;68:267-89.
2. Schneider LS. Pharmacologic management of psychosis in dementia. J Clin Psychiatry 1999;60(Suppl 8):54-60.
3. Tariot PN. Treatment of agitation in dementia. J Clin Psychiatry 1999;60(Suppl 8):11-20.
4. Levy ML, Cummings JL, Kahn-Rose R. Neuropsychiatric symptoms and cholinergic therapy for Alzheimer's disease. Gerontology 1999;45(Suppl 1):15-22.
5. Casey DE. Side effect profiles of new antipsychotic agents. J Clin Psychiatry 1996;57(Suppl 11):40-5.
6. Zayas EM, Grossberg GT. The treatment of psychosis in late life. J Clin Psychiatry 1998;59(Suppl 1):5-10.
7. Rogers SL, Doody RS, Mohs RC, et al. Donepezil improves cognition and global function in Alzheimer disease: a 15-week, double-blind, placebo-controlled study. Donepezil Study Group. Arch Intern Med 1998;158(9):1021-31.
8. Wengel SP, Roccaforte WH, Burke WJ. Donepezil improves symptoms of delirium in dementia: implications for future research. J Geriatr Psychiatry Neurol 1998;11(3):159-61.
9. Mega MS, Masterman DM, O'Connor SM, et al. The spectrum of behavioral responses to cholinesterase inhibitor therapy in Alzheimer disease. Arch Neurol 1999;56:1388-93.
10. Burt T. Donepezil and related cholinesterase inhibitors as mood and behavioral controlling agents. Curr Psychiatry Rep 2000;2:473-8.
11. Burke WJ, Roccaforte WH, Wengel SP. Treating visual hallucinations with donepezil. Am J Psychiatry 1999;156:1117-8.
12. Rogers SL, Friedhoff LT. The efficacy and safety of donepezil in patients with Alzheimer's disease: results of a US Multicentre, Randomized, Double-Blind, Placebo- Controlled Trial. The Donepezil Study Group. Dementia 1996;7(6):293-303.
13. Burns A, Rossor M, Hecker J, et al. The effects of donepezil in Alzheimer's disease - results from a multinational trial. Dement Geriatr Cogn Disord 1999;10:237-44.
14. Dooley M, Lamb HM. Donepezil: a review of its use in Alzheimer's disease. Drugs Aging 2000;16:199-226.
15. Cummings JL, Gorman DG, Shapira J. Physostigmine ameliorates the delusions of Alzheimer's disease. Biol Psychiatry 1993;33:536-41.
16. Kaufer DI, Cummings JL, Christine D. Effect of tacrine on behavioral symptoms in Alzheimer's disease: an open-label study. J Geriatr Psychiatry Neurol 1996;9:1-6.
17. McKeith I, Del Ser T, Spano P, et al. Efficacy of rivastigmine in dementia with Lewy bodies: a randomised, double-blind, placebo-controlled international study. Lancet 2000;356(9247):2031-6.
18. Bergman J, Lerner V. Successful use of donepezil for the treatment of psychotic symptoms in patients with Parkinson's disease. Clin Neuropharmacol 2002;25:107-10.
19. Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res 1975;12:189-98.
20. Reisberg B, Ferris SH, de Leon MJ, et al. Global Deterioration Scale (GDS). Psychopharmacol Bull 1988;24:661-3.
21. Pollock BG, Mulsant BH, Rosen J, et al. Comparison of citalopram, perphenazine, and placebo for the acute treatment of psychosis and behavioral disturbances in hospitalized, demented patients. Am J Psychiatry 2002;159:460-5.
22. Sweet RA, Pollock BG, Mulsant BH, et al. Pharmacologic profile of perphenazine's metabolites. J Clin Psychopharmacol 2000;20:181-7.
23. Kay S, Opler L, Fiszbein A. Positive and Negative Syndrome Scale (PANSS) Manual. North Tonawanda, NY: Multi-Health Systems; 1986.
24. Guy W. ECDEU Assessment Manual for Psychopharmacology, revised. Washington, DC: US Department of Health, Education and Welfare; 1976.

    .

ELIGIBILITY:
Inclusion Criteria:

* age: 65-90
* DSM-IV diagnosis of Alzheimer's type dementia
* inclusion of psychotic symptoms such as: hallucinations and delusions, aggression/agitation, irritability and disinhibition calling for adminstration of antipsychotic drugs
* duration of psychotic symptoms of at least 2 weeks before start of treatment
* lack of improvement of psychotic symptoms during perphenazine treatment for at least 3 weeks

Exclusion Criteria:

* vascular demential
* concurrent Axis I DSM-IV diagnosis (delirium, schizophrenia, delusional disorder and affective disorders)
* significant medical illness (cardiovascular, liver, renal, edocrinal, B12 or folic acid deficience and neurological illnesses)
* drug or alcohol addiction

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)

PRIMARY OUTCOMES:
Possitive and Negative Syndrome Scale
Clinical Global Impression

CONTACTS AND LOCATIONS:
Overall Officials: Valdimir Lerner, MD, PhD, Principal Investigator — Ben-Gurion University of the Negev; Tzvi Dwolatzky, MD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Beersheva Mental Health Center, Beersheva, Israel